CLINICAL TRIAL: NCT05500365
Title: Development and Clinical Validation of an In Silico Pace Mapping Approach Utilising Implanted Device Electrograms to Accurately Guide Ventricular Tachycardia Ablation
Brief Title: In Silico Pace Mapping To Optimise Ventricular Tachycardia Ablation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: v1.0
Record Dates: First submitted 2022-04-04; First posted 2022-08-15 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-08

CONDITIONS: Ventricular Tachycardia
Keywords: Catheter Ablation; Pace Mapping
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation therapy — Pace mapping procedure performed during catheter ablation therapy

SUMMARY:
People who suffer from incessant cardiac arrhythmias receive a small electrical device implanted into their chest that automatically senses when the heart beats arrhythmically and applies electrical pulse to re-establish normal activity. However, if problems persist, people can have an operation called catheter ablation therapy, which involves 'burning' small areas of the heart tissue in order to permanently disrupt the problematic electrical pathways driving these arrhythmias.

However, procedure times and complication rates are high, whist success rates are punitively low (~50% success), largely due to the significant challenge clinicians face in identifying the ideal 'target' to ablate within the patient's heart. In this project, the investigators aim to develop, and clinically validate, an in silico tool that reconstructs a personalised computational model of a patient's heart using advanced MRI data, upon which a virtual 'mapping' procedure is then performed in order to identify (in the model) the optimal ablation target. This pre-procedural planning tool utilises stored information about the patient's specific arrhythmia from their implanted device, ensuring optimal targets are selected. The approach aims to reduce procedure times whilst increasing their safety, and ensure significantly increased long-term effectiveness of these invasive ablation procedures, increasing survival rates and quality-of-life.

This study is concerned with the clinical arm of the study, specifically, in the collection of data from patients in order to (retrospectively) validate the computational model. The model itself will not be applied or used to treat these patients.

DETAILED DESCRIPTION:
Catheter ablation of ventricular tachycardia (VT) most frequently requires the identification of exit sites of slow-conducting diastolic isthmuses associated with infarcted tissue which are critical to sustain the reentrant arrhythmia. Pace mapping is a technique that identifies exit sites by matching the recorded 12-lead electrocardiogram (ECG) QRS of catheter-paced beats at different myocardial locations with the QRS of the clinical VT. When a high correlation between QRS morphologies is found, it is believed that the paced-beat lies at the VT exit site, helping guide the ablation. Procedures thus involve methodologically moving the catheter to multiple (accessible) locations to produce a pace map. Unfortunately the procedure is inherently limited due to the following reasons:

i) Surface maps - Most often, pacing sites are limited to the endocardium (where catheter access is easiest). Consequently, identification of VTs with an intramural or epicardial substrate can be challenging, with mis-leading and/or difficult to interpret pace maps being obtained.

ii) Low Resolution - Due to time-pressures and practical difficulties in catheter manipulation, pace map sites are often sparsely located (typically 40-60 separate sites). In complex structural VTs, with multiple possible anatomical circuits through the scar, it is often challenging to accurately identify from the map the relevant isthmus exit site responsible for the presenting clinical VT.

iii) VT Induction - Pace mapping usually necessitates VT induction during the procedure, which is time-consuming and carries inherent risk (~80% of induced VTs in ischemic heart disease (IHD) are either non-sustained or not haemodynamically tolerated), but induction of the exact clinical VT itself is often challenging.

A non-invasive, pre-procedural approach that is capable of generating accurate, high-resolution 3-dimensional personalised pace maps that correlate with the presenting clinical VT without the need for VT induction would thus revolutionise VT ablation planning, guidance, safety and efficacy.

Two recent studies have demonstrated the utility of performing a pace map based on comparison to stored implanted cardioverter defibrillator (ICD) electrograms (EGMs) of the clinical VT. The first study initially demonstrated that stored ICD EGMs allow differentiation of the clinical VT from other VTs, and their subsequent use in pace mapping may be useful for identifying the VT exit site. More recently, it has been prospectively shown that pace mapping of non-inducible clinical VTs based on ICD EGMs is feasible and resulted in higher freedom from recurrent VT, compared to targeting only inducible VTs.

The investigators have recently published a pipeline for creating a patient-specific image-based whole torso-cardiac model to perform virtual ('in silico') pace mapping. The approach creates a high-resolution 3D pace map that successfully identifies the exit site of an induced (simulated) VT within the same model, using both simulated 12-lead ECG and ICD EGM data derived from the simulated VT episode. Here, it was demonstrated: 1) the importance of creating a dense, fully transmural (3D) pace map to allow differentiation of epicardial vs endocardial substrates; 2) that accuracy of exit site identification could be enhanced by considering multiple EGM sensing vectors, e.g. from multipolar cardiac resynchronisation devices (CRT-D) with additional epicardial electrodes. Developed on simulated data, this workflow now requires full validation with clinical data from ablation patients, as proposed here, and refinement of methodological algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 99 years
* Ability to provide informed consent to participate and willing to comply with the clinical investigation plan and follow-up schedule.
* Ventricular tachycardia secondary to ischemic heart disease clinically indicated for catheter ablation therapy
* Cardiac implanted electronic device in situ

Exclusion Criteria:

1. Standard contra-indications to VT ablation
2. Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
3. Contra-indication to contrast agent for Cardiac MRI scan
4. Implanted device that is not MRI-conditional

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Ischemic cardiomyopathy suffering from refractory ventricular tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Performance of in silico derived pace map | At the time of the procedure.
  The primary outcome measure will be the geometrical distance between the exit site (site of highest correlation) identified from the in silico pace map (created from the collected patient data) and the actual pace map derived from the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Rinaldi, MD, Principal Investigator — St Thomas' Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoshida K, Liu TY, Scott C, Hero A, Yokokawa M, Gupta S, Good E, Morady F, Bogun F. The value of defibrillator electrograms for recognition of clinical ventricular tachycardias and for pace mapping of post-infarction ventricular tachycardia. J Am Coll Cardiol. 2010 Sep 14;56(12):969-79. doi: 10.1016/j.jacc.2010.04.043. PMID 20828650
- [Background] Yokokawa M, Kim HM, Sharaf Dabbagh G, Siontis KC, Lathkar-Pradhan S, Jongnarangsin K, Latchamsetty R, Morady F, Bogun F. Targeting Noninducible Clinical Ventricular Tachycardias in Patients With Prior Myocardial Infarctions Based on Stored Electrograms. Circ Arrhythm Electrophysiol. 2019 Jul;12(7):e006978. doi: 10.1161/CIRCEP.118.006978. Epub 2019 Jun 20. PMID 31216885
- [Result] Monaci S, Strocchi M, Rodero C, Gillette K, Whitaker J, Rajani R, Rinaldi CA, O'Neill M, Plank G, King A, Bishop MJ. In-silico pace-mapping using a detailed whole torso model and implanted electronic device electrograms for more efficient ablation planning. Comput Biol Med. 2020 Oct;125:104005. doi: 10.1016/j.compbiomed.2020.104005. Epub 2020 Sep 17. PMID 32971325